CLINICAL TRIAL: NCT03605719
Title: PD1 Blockade and Oncolytic Virus in Relapsed Multiple Myeloma
Brief Title: Dexamethasone, Carfilzomib, & Nivolumab With Pelareorep for Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Bristol-Myers Squibb (Industry); Oncolytics Biotech (Industry); University of Utah (Other); City of Hope Medical Center (Other); Phylogeny (Unknown); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Craig Hofmeister, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00104234; NCI-2018-01217 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4398-18 (Other: Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Recurrent Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Dexamethasone; Calcium Dobesilate; Nivolumab; reolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Patients receive dexamethasone IV on days 1, 2, 8, 9, 15, and 16, carfilzomib IV over 30 minutes on days 1, 2, 8, 9, 15, and 16, and nivolumab IV over 30 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Biological: Nivolumab
- Arm 2 (Experimental): Patients receive dexamethasone IV on days 1, 2, 8, 9, 15, and 16, pelareorep IV on days 1, 2, 8, 9, 15, and 16, carfilzomib IV over 30 minutes on days 1, 2, 8, 9, 15, and 16, and nivolumab IV over 30 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Biological: Nivolumab; Biological: Pelareorep
- Arm 3 (expansion) (Experimental): Patients receive dexamethasone IV on days 1, 2, 8, 9, 15, and 16, pelareorep IV on days 1, 2, 8, 9, 15, and 16, carfilzomib IV over 30 minutes on days 1, 2, 8, 9, 15, and 16, and nivolumab IV over 30 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Biological: Nivolumab; Biological: Pelareorep

INTERVENTIONS:
Drug: Carfilzomib — Given IV
  Other Names: Kyprolis; PR-171
Drug: Dexamethasone — Given IV
  Other Names: Decadron; Hexadrol; Ozurdex
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Biological: Pelareorep — Given IV
  Other Names: Reolysin; Wild-type Reovirus
  Arms: Arm 2; Arm 3 (expansion)

SUMMARY:
This phase I trial studies the side effects and best dose of wild-type reovirus (pelareorep) when given together with dexamethasone, carfilzomib, and nivolumab in treating patients with multiple myeloma that has come back (relapsed). Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer and may interfere with the ability of tumor cells to grow and spread. A virus, called pelareorep, which has been changed in a certain way, may be able to kill tumor cells without damaging normal cells. Giving dexamethasone, carfilzomib, and nivolumab with pelareorep may work better in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify maximum tolerated dose of pelareorep in combination with other antineoplastic agents.

II. Identify whether the combination of carfilzomib and nivolumab lead to a safety profile different than what has been reported with either agent independently.

SECONDARY OBJECTIVES:

I. Assess the relative roles of immune-mediated and direct cytotoxic myeloma cell killing.

II. Understand the clinical benefit of nivolumab in programmed death-ligand 1 (PD-L1) positive multiple myeloma (MM) cells.

OUTLINE: This is a dose-escalation study of pelareorep. Patients are assigned to 1 of 3 arms.

ARM 1: Patients receive dexamethasone intravenously (IV) on days 1, 2, 8, 9, 15, and 16, carfilzomib IV over 30 minutes on days 1, 2, 8, 9, 15, and 16, and nivolumab IV over 30 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM 2: Patients receive dexamethasone IV on days 1, 2, 8, 9, 15, and 16, pelareorep IV on days 1, 2, 8, 9, 15, and 16, carfilzomib IV over 30 minutes on days 1, 2, 8, 9, 15, and 16, and nivolumab IV over 30 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM 3 (expansion cohort): Patients receive dexamethasone IV on days 1, 2, 8, 9, 15, and 16, pelareorep IV on days 1, 2, 8, 9, 15, and 16, carfilzomib IV over 30 minutes on days 1, 2, 8, 9, 15, and 16, and nivolumab IV over 30 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for a minimum of 4 weeks once off treatment or at least 100 days after the last nivolumab dose, then every 6 months after.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have multiple myeloma that fits or did fit International Myeloma Working Group (IMWG) diagnostic criteria
* In arm 3 but not for arms 1 or 2, patients must have measurable disease defined as any of the following:

  * Serum monoclonal protein ≥ 0.5 g/dL by protein electrophoresis
  * ≥ 200 mg of monoclonal protein in the urine on screening 24-hour electrophoresis
  * If no m-spike is present, involved serum immunoglobulin free light chain ≥ 100 mg/L AND an abnormal serum light chain ratio (< 0.26 or > 1.65)
* Progressive disease or clinical relapse at the time of study entry as defined by IMWG
* Arm ONE only: Patients must be carfilzomib naive and have received ≥ 2 prior lines of therapy and must have included an IMiD, proteasome inhibitor, and anti-cluster of differentiation 38 (CD38) antibody as defined below

  * IMiD exposure: At least 1 cycle of prior treatment unless stopped due to intolerance
  * CD38 antibody exposure: At least 4 doses unless stopped due to intolerance
  * Proteasome inhibitor exposed: At least 1 cycle of prior treatment unless stopped due to intolerance
* Arm TWO and THREE only: Patients must have received ≥ 3 prior lines of therapy and must have included an immunomodulatory imide drug (IMiD), proteasome inhibitor, and anti-CD38 antibody as above along with evidence of proteasome inhibitor resistance defined as less than or equal to stable disease with prior treatment with a proteasome inhibitor containing regimen at moderate doses defined as carfilzomib 27+ mg/m²/week (wk), bortezomib 1.3+ mg/m²/wk subcutaneously (SQ) or IV, or ixazomib 3+ mg/wk orally (PO)
* Both men and women of all races and ethnic groups are eligible for this study
* Eastern Cooperative Oncology Group (ECOG) performance status < 2 (Karnofsky > 60%) is required for eligibility. Those patients with lower performance status based solely on bone pain secondary to multiple myeloma are eligible
* Prior autologous and/or allogeneic transplant is permitted although transplant must have occurred greater than 90 days prior to registration
* Absolute neutrophil count (ANC) > 1000/µL for at least one week prior to screening
* Platelet count ≥ 70,000 and platelet transfusion independent for one week prior to screening (platelets allowed to be down to 50,000 if > 50% plasma cells on screening aspirate or core biopsy)
* Estimated creatinine clearance ≥ 30 mL/min as defined by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) or Cockcroft-Gault
* Total bilirubin < 1.5 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3x the institutional upper limit of normal
* Left ventricular ejection fraction ≥ 40%
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test prior to starting therapy. The effects of pelareorep and nivolumab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Female of childbearing potential (FCBP) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* The patient must be willing to comply with fertility requirements as below:

  * Male patients must agree to use an adequate method of contraception for the duration of the study and for 7 months afterwards
  * Female patients must be either postmenopausal, free from menses ≥ 2 years, surgically sterilized, willing to use two adequate barrier methods of contraception to prevent pregnancy, or agree to abstain from heterosexual activity starting with screening and for 5 months after last treatment in all patients
  * Patients must agree not to donate blood, sperm/ova while taking protocol therapy and for at least 7 months after stopping treatment (for males) and 5 months after stopping treatment (for females)
* Ability to understand and the willingness to sign a written informed consent document
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial

Exclusion Criteria:

* Known human immunodeficiency virus (HIV) infection or active hepatitis B or C due to risk of viral infectivity of pelareorep
* Known pulmonary hypertension
* Patients who are receiving any other anti-myeloma investigational agents
* Polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, skin changes (POEMS) syndrome, primary amyloidosis (AL amyloidosis), and Waldenstrom macroglobulinemia
* Patients who have had anti-myeloma treatment, radiotherapy, plasmapheresis, or major surgery (as defined by the investigator) within 2 weeks prior to cycle 1 day 1 of the study. Patients may be receiving concomitant therapy with bisphosphonates and low dose corticosteroids (e.g., prednisone up to but no more than 10 mg by mouth daily or its equivalent) for symptom management and comorbid conditions
* Uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, myocardial infarction in the preceding 6 months, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because protocol therapy has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to protocol treatment of the mother, breastfeeding should be discontinued

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) of 4-drug regimen evaluated according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) | Up to 28 days after cycle 1 start
  A DLT is defined as one of the following toxicities:
  * Grade 4 neutropenia (absolute neutrophil count [ANC] < 500/µL) lasting 5 days or more.
  * Grade 3 to 4 thrombocytopenia associated with bleeding requiring platelet transfusion
  * Cardiac dysfunction: Grade > 3 left ventricular systolic dysfunction or grade > 2 myocarditis
  * Any grade 3-4 treatment-emergent non-hematologic adverse event (AE) clearly unrelated to the underlying disease and considered to be at least possibly related to protocol therapy
Maximum tolerated dose (MTD) of 4-drug regimen | Up to 28 days after cycle 1 start
  The Escalation with Overdose Control (EWOC) design will be used to identify the MTD.
DLT of 3-drug regimen evaluated according to NCI CTCAE version 5.0 | Up to 28 days after cycle 1 start
  A DLT is defined as one of the following toxicities:
  * Grade 4 neutropenia (absolute neutrophil count [ANC] < 500/µL) lasting 5 days or more.
  * Grade 3 to 4 thrombocytopenia associated with bleeding requiring platelet transfusion
  * Cardiac dysfunction: Grade > 3 left ventricular systolic dysfunction or grade > 2 myocarditis
  * Any grade 3-4 treatment-emergent non-hematologic adverse event (AE) clearly unrelated to the underlying disease and considered to be at least possibly related to protocol therapy

SECONDARY OUTCOMES:
Time to progression | From start of protocol therapy up to 3 years
  Defined as the time from start of protocol therapy until the criteria for disease progression are met. Patients who are either lost to follow-up, die or who begin alternative treatments prior to progression, will have their data censored as of the date considered to be lost to follow-up, date of death, or the first day of alternative therapy.
Progression-free survival | From start of protocol therapy up to 3 years
  Defined as the time from start of protocol therapy to disease progression or death from any cause, censoring patients without an event at time of last clinical assessment.
Overall survival | From start of protocol therapy up to 3 years
  Defined as the time from start of protocol therapy to death, censoring patients who are alive at last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hofmeister, MD, MPH, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

DOCUMENTS (1):
  • Informed Consent Form (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT03605719/ICF_000.pdf